CLINICAL TRIAL: NCT02088099
Title: The CONNECT Trial: A Randomized Pragmatic Clinical Trial Measuring the Effectiveness of a Remotely Provided Complex Brain Rehabilitation Intervention in Improving Participation Outcomes of Individuals With TBI, Their Families, and Local Primary Providers
Brief Title: Mayo Clinic Traumatic Brain Injury Model System Center: The CONNECT Trial
Acronym: CONNECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Minnesota Department of Health (Other Government); Iowa Department of Public Health (Unknown); Rapid City Regional Hospital, Inc (Other); Altru Health System (Other)
Responsible Party: Principal Investigator, Allen Brown, PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12-008525; NIDILRR (Other Grant/Funding Number: H133A120026)
Record Dates: First submitted 2014-03-12; First posted 2014-03-14 (Estimated); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic brain injury; Telehealth; ehealth; Mobile Health; social participation; patient participation; consumer participation; Patient Outcome Assessment
MeSH Terms: conditions — Brain Injuries, Traumatic; Patient Participation | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Complex clinical intervention (Experimental)
  Interventions: Other: Complex clinical intervention
- Treatment as usual (Active Comparator)
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Other: Complex clinical intervention — The complex intervention in CONNECT will be tested in 3 target populations: (1) Individuals hospitalized for TBI; (2) their family members; (3) their local health care providers. All intervention components will be delivered remotely: there will be no face-to-face interaction with the research subjects. The complex intervention tested in CONNECT is comprised of the clinical direction and advice to local providers, educational, and supportive services of the Mayo Brain Rehabilitation Clinic (BRC). The specific communication modes used to interact with individual study subjects, and the specific clinical and educational support services that are provided to an individual subject by these modes, will be determined by clinical need, individual preference, and technological capacity.
  Arms: Complex clinical intervention
Other: Treatment as usual — Participants in this arm will receive, experience, or provide the care that is usual and customary in their communities.
  Arms: Treatment as usual

SUMMARY:
Mayo Clinic has been funded by the National Institute on Disability Independent Living & Rehabilitation Research (NIDILRR) as a Traumatic Brain Injury (TBI) Model System Center continuously since 1998. We have successfully competed for this funding because we consistently produce high quality research and because we provide comprehensive team-based rehabilitation services to people with TBI and their families over the continuum of care that is associated with superior outcomes.

Lack of access to specialized TBI care is the most common need identified by individuals after they are hospitalized for TBI. The upper Midwest has some of the highest populations of rural dwellers, the elderly, and Native Americans, all of whom have a high risk for TBI and are more likely to have limited access to rehabilitation services after acute care. Explosive advances in communication technology have brought tele-medicine to the forefront of health care. The CONNECT trial will test the effectiveness of using modern technologies - such as phone consultation and other telehealth communication systems - to deliver specialized brain rehabilitation resources remotely to patients and providers in the upper Midwest. The groups targeted by the CONNECT trial are:

* Individuals recently hospitalized with TBI;
* Their families;
* Their local health care and other providers (primary care providers, psychologists, therapists, social service providers, job counselors).

The CONNECT trial is the first study of this scope - in 4 upper Midwest states (MN, IA, ND, and SD), 3 health systems (Mayo Clinic, Altru Health System in ND, Regional Health in SD), and 2 state Departments of Health (IA, MN) - using electronic technology to see if outcome can be improved by providing care with no face-to-face contact. The trial will study whether outcomes over three years are different in the group receiving this remotely provided model of care compared to a matched group that receives usual care in their communities.

The desired long term outcome of this study is to increase our capacity to provide care and to reduce barriers to accessing specialized TBI rehabilitation services faced by individuals with TBI and their families.

DETAILED DESCRIPTION:
MAYO CLINIC TRAUMATIC BRAIN INJURY MODEL SYSTEM CENTER:

The CONNECT Trial

Connecting the upper Midwest traumatic brain injury community to Mayo Clinic and each other: providing research evidence of effectiveness for remote support and care coordination

Problem: Traumatic brain injury (TBI) is a common injury and cause of disability in the US, yet there are few medical practices specialized in treating post-acute and chronic impairment, activity limitations, and restrictions to community participation and employment that often result from TBI. This is of particular concern in rural areas, among the elderly, and in the Native American population.

Gap in knowledge: Evidence exists for the effectiveness of care provided by multi-discipline clinical rehabilitation teams in treating the complex medical, cognitive, and psychosocial sequelae of TBI and improving outcome. Some evidence exists for the effectiveness of remotely provided services, such as cognitive rehabilitation. Mayo Clinic's specialty brain rehabilitation practice has experience with assembling treatment teams in remote communities and providing clinical guidance, with positive anecdotal reports of effectiveness. However, there currently exists no research evidence indicating such intervention is superior to treatment as usual (TAU).

Research design: In collaboration with the Departments of Health in Iowa and Minnesota, Regional Health in South Dakota, and Altru Health System in North Dakota, Mayo Clinic's TBI Model System Center will recruit 500 individuals discharged from the hospital over a year's time with an ICD-9/10 diagnosis of TBI. Subjects will be randomized by demographic and urban/rural status into two groups: an intervention group and a TAU group. Subjects in the intervention group will be remotely interviewed and evaluated by Mayo's clinical team. Their rehabilitation needs will be assessed and connections made to local health care and community providers who will receive TBI-specific education and consultative support from Mayo's TBI Model System Center staff. The target populations who will be consented are: 1) individuals with TBI; 2) their family members or caregivers; and 3) their local care providers. All consented subjects will be followed regularly for up to 3 years. All available resources in an individual's community, and within Mayo's TBI Model System Center, will be used to: 1) CONNECT the coordinating team with subjects and their families; 2) CONNECT the coordinating team with local medical, rehabilitation and community providers; and 3) CONNECT individuals with TBI, their families, and local providers with each other. Patient and family education, long term support, care coordination and clinical advice will be provided to intervention group subjects, their families and local clinicians remotely via traditional, web based, and social media platforms. Subjects in the usual care group will receive the care they would normally receive in their respective communities (TAU). Clinical, demographic, subject-reported outcomes, medical economic estimates, and satisfaction/competence measures will occur at baseline, midpoint, and at study end. Primary outcome measures will include measures of impairment, activity limitations, and participation with a primary focus on outcomes related to independent living, employment, and quality of life. The hypothesis is that outcomes in the remotely coordinated intervention group will be superior to outcomes in the group that received TAU.

If study results support this hypothesis, a hub-based system of remotely coordinated brain rehabilitation care could be considered, using the TBI Model System Centers as test sites that could revolutionize the provision of medical care and post acute support for individuals with TBI and their families.

ELIGIBILITY:
Inclusion Criteria:

* English speaking individuals who are at least 18 years old
* Hospitalized for a minimum of 24 hours (no maximum) with TBI during the recruitment window in one of the following: 1) Hospital in state of Minnesota, 2) Hospital in state of Iowa, 3) Regional Health, 4) Altru Health System
* Individuals with TBI who have (or their LAR has) at least telephone communication technology

Exclusion Criteria:

* Non-English speaking individuals
* Individuals under a civil commitment order
* Individuals with TBI who are in coma or minimally conscious (not following commands)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 426 (Actual)
Dates: Start 2014-03; Primary Completion 2017-09 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change in Traumatic Brain Injury - Quality of Life (TBI-QOL) | At enrollment, at 6 months, and at 18 months
  TBI-QOL is a recently developed Computer Assisted Telephone Interview (CATI) tool that provides psychometrically sound and clinically relevant health-related patient-reported quality of life measurement specific to TBI. This scale is being used by the VA Research and Development Programs and will soon be a variable in the TBIMS National Database. TBI-QOL efficiently measures domains of depression, anxiety, fatigue and pain, using fewer items than scales measuring similar constructs. Responses for this scale will be obtained from subjects via a CATI.
Change in measure of patient impression of Telemedicine (TMP-Q) | At enrollment, at 6 months, and at 18 months
  Given that the entire complex intervention of this trial is delivered remotely, individual differences in its acceptance may influence outcome. The TMP-Q is a 17-item scale designed to assess impressions of the risks and benefits of home tele-care, and that has high levels of test-retest reliability and validity. Responses to a revised TMP-Q customized for the CONNECT trial will be obtained directly from subjects by phone interview or on-line via the protected and secure web-based CONNECT trial CareHubs site.
Change in Caregiver Appraisal Scale (CAS) | At enrollment, at 6 months, and at 18 months
  The CAS will be used only for family members or care givers to measure caregiver burden. It contains 4 measurable factors: Perceived Burden, Caregiver Satisfaction, Caregiver Idealogy and Caregiver Mastery. It includes 35 questions each measured on a 5-point Likert scale. The CAS has high internal consistency when used to study burden in those caring for individuals with TBI. Responses for this scale will be obtained from family members and caregivers via phone interview or on-line via the protected and secure web-based CONNECT trial CareHubs site.
Change in Clinical Satisfaction and Competency Rating (CSCR) | At enrollment, at 6 months, and at 18 months
  CSCR scales use a 5-point Likert method to measure satisfaction specific to individuals in each target population. They will be tested and refined in small groups of the target populations during Phase 1. The CSCR scale for individuals with TBI will focus on intervention quality, services, and progress. Satisfaction for family members will emphasize coping, communication, learning, and access. Questions to local providers will focus on their comfort, confidence, and competency in providing care to individuals with TBI. Responses for these scales will be obtained from individuals with TBI, their family members/caregivers, and their primary providers via phone interview or on-line via the protected and secure web-based CONNECT trial CareHubs site.

SECONDARY OUTCOMES:
Change in the Activity Measure for Post-Acute Care™ (AM-PAC™) | At enrollment, at 6 months, and at 18 months
  AM-PAC™ is a state-of-the-art outcome instrument that measures function in three domains: basic mobility, daily activities and applied cognition. The AM-PAC™ is used for quality improvement, outcomes monitoring, and research activities in inpatient and outpatient rehabilitation, home care, nursing homes and long-term acute care settings. The AM-PAC™ is appropriate for functional assessment in adults with a wide range of diagnoses and functional abilities. Patients will respond to AM-PAC™ test items using a computer-based version similar to the data collection forms loaded into Assessment Center. Research subjects will be sent a customized link to AM-PAC™ for each point of data collection (enrollment, 6 months, 18 months) and will complete data entry via this user-friendly system at their convenience, within established data collection windows, for example, +/- 1 month at 6 month data collection. Reminders will be sent as needed and short paper forms mailed to non-responders.
Change in self-reported use of health care and other community support services | Every 3 months after consenting until the end of study period at 18 months
  Every 3 months after consenting until the end of study period at 18 months, each consented individual with TBI or their LAR in both groups will be contacted by phone or on-line via the protected and secure web-based CONNECT trial CareHubs site to determine their self-reported use of health care and other community support services.

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Bergquist TF, Moessner AM, Mandrekar J, Ransom JE, Dernbach NL, Kendall KS, Brown AW. CONNECT: A pragmatic clinical trial testing a remotely provided linkage to service coordination after hospitalization for TBI. Brain Inj. 2022 Jan 28;36(2):147-155. doi: 10.1080/02699052.2022.2042601. Epub 2022 Feb 22. PMID 35192438